CLINICAL TRIAL: NCT04788498
Title: Laparoendoscopic Single-site Surgery Versus Conventional Multi-port Laparoscopy in Presumed Benign Ovarian Cystectomy: A Randomized Controlled Trial
Brief Title: Laparoscopic Single-site Surgery Versus Conventional Entry in Ovarian Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Nabil, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M D 34 / 2021
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cyst Benign

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoendoscpoic single site surgery LESS (Experimental): 35 patients undergoing laparoscopic ovarian cystectomy A SILS Port (Covidien®) with three access inlets will be inserted into the abdominal cavity using a Heaney clamp
  Interventions: Procedure: Laparoendoscpoic single site surgery LESS
- Conventional multiport laparoscopy (Active Comparator): 35 patients undergoing laparoscopic ovarian cystectomy It will be performed using a three-port system using a closed technique on the umbilicus, left and right lower quadrant area.
  Interventions: Procedure: Conventional multiport laparoscopy

INTERVENTIONS:
Procedure: Laparoendoscpoic single site surgery LESS — • A SILS Port (Covidien®) with three access inlets will be inserted into the abdominal cavity using a Heaney clamp
  Arms: Laparoendoscpoic single site surgery LESS
Procedure: Conventional multiport laparoscopy — • It will be performed using a three-port system using a closed technique on the umbilicus, left and right lower quadrant area.
  Arms: Conventional multiport laparoscopy

SUMMARY:
The aim of this work is to evaluate the postoperative consequences of laparoendoscopic single site surgery relative to conventional laparoscopy in presumed benign ovarian cyst.

The hypothesis is that single incision technique might offer advantages over the standard multi-port laparoscopy as potentially leading to less postoperative pain and improved cosmoses from a relatively hidden umbilical scar, as well as risk reduction of postoperative wound infection, hernia formation and elimination of multiple trocar site closure

ELIGIBILITY:
Inclusion Criteria:

* The patients are aged 18 to 45 years with BMI < 35 kg/m2 and that they exhibit a surgical indication for a presumed benign ovarian pathology (PBOP) according to RCOG Guideline no. 62. 2011:

  * simple ovarian cysts >7cm and <15cm.
  * Persistent simple cyst for more than 3 months.
  * Symptomatic patients with complicated cyst (e.g. hemorrhagic cyst, torsion, etc)

Exclusion Criteria:

* • Previous midline laparotomies as suspected massive adhesions affecting intraoperative maneuvers and time.

  * Chronic pelvic pain, endometriosis or pelvic inflammatory diseases will be excluded to avoid pelvic adhesions and bias in the quantification of postoperative pain.
  * Do not possess a native umbilicus giving difficult access to single port.
  * The 'risk of malignancy index' (RMI) should be used to exclude those women at greater risk of malignancy. Using an RMI cut-off of 200, a sensitivity of 70% and specificity of 90% can be achieved. if features suggestive of malignancy are encountered, a gynecological oncologist should be consulted regarding further evaluation and staging.
  * Benign teratomas for the difficulty of extraction after removal that affects the intraoperative maneuvers and time.
  * Contraindication to any laparoscopy like any medical condition worsened by pneumoperitoneum or the Trendelenburg position.
  * Contraindication to general anesthesia as all laparoscopic procedures are done under GA.
  * Contraindication to non-steroidal anti-inflammatories, paracetamol, or tramadol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | at 24 hours ± 2 hour after the intervention
  The pain will be assessed by a numeric rating scale of 0-10

SECONDARY OUTCOMES:
Operative time | intraoperative
  the time between the start of the incision up to the cutaneous closing of the trocar orifices
the need for conversion to laparotomy | intraoperative
  the need for conversion to laparotomy
the need to add an additional trocar | intraoperative
  the need to add an additional trocar

IPD SHARING:
Plan to Share IPD: No